CLINICAL TRIAL: NCT04866771
Title: Remotely Supervised Transcranial Direct Current Stimulation for Slowing Disease Progression in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Remotely Supervised tDCS for Slowing ALS Disease Progression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Sangeetha Madhavan, Associate Professor, Physical Therapy, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-0097
Record Dates: First submitted 2021-03-30; First posted 2021-04-30 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Direct Current Stimulation (tDCS) (Experimental): Facilitatory transcranial direct current stimulation (tDCS)
  Interventions: Other: Transcranial Direct Current Stimulation (tDCS)
- Delayed-Start Transcranial Direct Current Stimulation (tDCS) Control Group (Sham Comparator): Sham tDCS followed by a switch to anodal tDCS.
  Interventions: Other: Sham tDCS + anodal tDCS

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation (tDCS) — Noninvasive brain stimulation
  Other Names: Soterix Medical 1X1 tDCS mini-CT Stimulator
  Arms: Transcranial Direct Current Stimulation (tDCS)
Other: Sham tDCS + anodal tDCS — Fake noninvasive brain stimulation or anodal noninvasive brain stimulation
  Other Names: Soterix Medical 1X1 tDCS mini-CT Stimulator
  Arms: Delayed-Start Transcranial Direct Current Stimulation (tDCS) Control Group

SUMMARY:
Most ALS care is centered on patient support and symptom management, making rehabilitation an integral aspect for slowing disease progression, prolonging life span, and increasing quality of life. Brain stimulation has been increasingly explored as a promising neuromodulatory tool to prime motor function in several neurological disorders. We propose a novel mechanism using remotely supervised brain stimulation to preserve motor function in individuals with ALS. This project will also aim to explore the effectiveness of brain stimulation on upper and lower motor neuron mechanisms in individuals with ALS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, probable, or definite amyotrophic lateral sclerosis according to El Escorial revised criteria
* Spinal onset ALS with initial weakness in the upper or lower extremity.
* Diagnosed with ALS within the past 5 years
* 1-2 point change in pre-slope of the ALSFRS-R at time of enrollment (ratio of drop in score from 48 to the duration in months from onset of weakness)
* Score ≥ 2 for "swallowing" of the ALSFRS-R
* Score ≥ 2 for "walking" of the ALSFRS-R
* Able to provide informed consent
* Stable dose of riluzole, edaravone, AMX0035 (Relyvrio) or no medications
* Availability of a caregiver for remote administration of tDCS

Exclusion Criteria:

* Subject has bulbar onset ALS
* Any neurological diagnosis other than ALS
* Psychiatric disorders
* Any other concomitant disease that affects prognosis of ALS inclusive of systemic disease, cardiovascular disease, hepatic or renal disorder
* Tracheostomal or noninvasive ventilation for more than 12 hours per day
* Enrollment in an on-going ALS pharmaceutical trial
* Subject plans on moving within 6 months.

TMS Exclusion Criteria:

* Implanted cardiac pacemaker
* Metal implants in the head or face
* Unexplained, recurring headaches
* History of seizures or epilepsy
* Currently under medication that could increase motor excitability and lower seizure threshold
* Skull abnormalities or fractures
* Concussion within the last 6 months
* Currently pregnant
* tDCS Exclusion Criteria:
* Skin hypersensitivity
* History of contact dermatitis
* History of allodynia and/or hyperalgesia
* Any other skin or scalp condition that could be aggravated by tDCS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Madhavan, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Brain Plasticity Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madhavan S, Deshmukh S, Cummings M, Doshi A, Rezania K, Freels S, Sawa G. Home-Based Tele-tDCS in Amyotrophic Lateral Sclerosis: Feasibility, Safety, and Preliminary Efficacy. Ann Clin Transl Neurol. 2025 May;12(5):1022-1033. doi: 10.1002/acn3.70038. Epub 2025 Mar 24. PMID 40125702

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 70 individuals were assessed for eligibility. Of these, 56 were excluded prior to randomization: 48 did not meet eligibility criteria and 8 declined to participate or were unable to commit due to logistical reasons. Fourteen participants were randomized (7 to the intervention group and 7 to the delayed-start group). All eligibility assessments and consent were conducted remotely or in person before randomization.
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Delayed-Start Transcranial Direct Current Stimulation (tDCS) Control Group
Started | 7 | 7
Completed | 7 | 3
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Delayed-Start Transcranial Direct Current Stimulation (tDCS) Control Group | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (9) | 55 (10) | 54 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Revised ALS Functioning Rating Scale (ALSFRS-R)
Description: This questionnaire evaluates function over time and disease progression in ALS patients with questions related to daily activities such as speech, swallowing, walking, etc. Scores range between 0-48 with higher scores corresponding to more function being retained.
Time Frame: Change from baseline to immediately after training and baseline to 3 months follow up.
Population: Analyses were conducted on an intent-to-treat basis, including all randomized participants who received at least one session. Missing data were handled using the last observation carried forward (LOCF) approach.
Measure: Mean (Standard Error); unit: Change score on ALSFRS-R
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Delayed-Start Transcranial Direct Current Stimulation (tDCS) Control Group
Number analyzed (Participants) | 7 | 7
Change score on ALSFRS-R
  Pre to Post | -1 (1.06) | -7.1 (1.56)
  Pre to 3 month follow up | -3.2 (2) | -7.1 (1.56)

2. Secondary Outcome: Gait Speed
Description: Self-selected will be measured as the average walking speed from 2 trials of the 10-m walk test (10MWT).
Time Frame: Change from baseline to immediately after training
Population: Gait speed data were collected for participants who were able to complete the 10MWT. Participants (n=6) who were non-ambulatory and could not perform the test at baseline or follow-up, and were therefore excluded from this analysis. Participants who withdrew from the study or did not complete the intervention are also not included in the analyses
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Delayed-Start Transcranial Direct Current Stimulation (tDCS) Control Group
Number analyzed (Participants) | 6 | 2
m/s | -0.11 (0.1) | -0.30 (0.08)

3. Secondary Outcome: Ankle Motor Control
Description: The participant will track a computer-generated sinusoidal target with ankle dorsiflexion and plantarflexion in a custom-built ankle-tracking device. Accuracy of tracking the target with ankle motion will be calculated.
Time Frame: Change from baseline to immediately after training and baseline to 3 months follow up.
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Quality of Life With EuroQol-5D (EQ-5D)
Description: Quality of life will be measured with the EuroQol-5D (EQ-5D), a questionnaire with questions designed to assess aspects of quality of life.
Time Frame: Change from baseline to immediately after training and baseline to 3 months follow up.
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: EuroQual-Visual Analog Scale (EQ-VAS)
Description: Quality of life will be measured using a visual analog scale with endpoints labeled, 'The best health you can imagine' and 'the worst health you can imagine' in response to questions related to aspects of quality of life. Scores range from 0 to 100, with higher values indicating better self-rated health status."
Time Frame: Change from baseline to immediately after training
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Fatigue Severity Scale
Description: 9-item scale measuring severity of fatigue and its effect on participant's daily activities and lifestyle with higher scores representing more fatigue and fatigue playing a larger role in daily activities. Minimum score = 0 and maximum score = 63.
Time Frame: Change from baseline to immediately after training.
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Upper and Lower Motor Neuron Mechanisms Using Transcranial Magnetic Stimulation (TMS)
Description: Upper and lower motor neuron mechanisms of the tibialis anterior will be measured using single pulse transcranial magnetic stimulation (TMS). Measures may include motor evoked potential (MEP) amplitude, latency, and/or cortical silent period.
Time Frame: Change from baseline to immediately after training and baseline to 3 months follow up.
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: Upper and Lower Motor Neuron Mechanisms Using Peripheral Nerve Stimulation (PNS)
Description: Upper and lower motor neuron mechanisms in ALS will also be assessed using peripheral nerve stimulation at either the knee or the elbow.
Time Frame: Change from baseline to immediately after training and baseline to 3 months follow up.
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: 24 weeks during intervention and 3-month follow-up period (total of ~36 weeks)
Description: Adverse events were monitored during each remotely supervised session using a structured questionnaire. Participants rated local and systemic symptoms (e.g., itching, tingling, redness) on a 0-4 scale. Definitions of adverse and serious adverse events aligned with ClinicalTrials.gov guidelines.
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Delayed-Start Transcranial Direct Current Stimulation (tDCS) Control Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transcranial Direct Current Stimulation (tDCS) (N=7) | Delayed-Start Transcranial Direct Current Stimulation (tDCS) Control Group (N=7)
Itching (Skin and subcutaneous tissue disorders) | 5 | 3
Tingling (Skin and subcutaneous tissue disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT04866771/Prot_SAP_000.pdf